CLINICAL TRIAL: NCT04413318
Title: A Cross-over Study to Compare Two Different Tracheal Cuff Pressure Monitoring Devices in a Pediatric Intensive Care Unit
Brief Title: Cuff Pressure Regulation Apparatus for Tracheal Intubation in Children
Acronym: CPRATIC-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: APHP190869; IDRCB: 2019-A02246-51 (Other: ANSM)
Record Dates: First submitted 2020-05-28; First posted 2020-06-02 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2020-05

CONDITIONS: Cuff Overinflation; Cuff Underinflation
Keywords: tracheal cuff pressure; pediatric critical care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- electronic device followed by pneumatic device (Experimental): Children receive continuous control of tracheal cuff pressure with the electronic device (VBM©) for 6-hours followed by continuous control of tracheal cuff pressure with the pneumatic device (Nosten©) for 6-hours.
  Interventions: Device: Electronic device (VBM©)
- pneumatic device followed by electronic device (Experimental): Children receive the reverse sequence (continuous control using the pneumatic device (Nosten©) for 6-hours followed by the electronic device (VBM©) for 6-hours
  Interventions: Device: Pneumatic device (Nosten©)

INTERVENTIONS:
Device: Electronic device (VBM©) — Continuous control of tracheal cuff pressure using an electronic device (VBM©) for 6-hours followed by continuous control using a pneumatic device (Nosten©) for 6-hours.
  Arms: electronic device followed by pneumatic device
Device: Pneumatic device (Nosten©) — Continuous control using a pneumatic device (Nosten©) for 6-hours followed by 6-hours of continuous control using an electronic device (VBM©).
  Arms: pneumatic device followed by electronic device

SUMMARY:
Despite the expert recommendation about rigorous monitoring of tracheal cuff pressure using a continuous or intermittent technique, cuff underinflation and overinflation are common increasing the risk of microinhalation and tracheal ischemia. All these complications are associated with high morbidity and mortality in ICU.

DETAILED DESCRIPTION:
In this study, the investigators will compare the duration of the period of under-inflation and over-inflation between electronic (VBM©) and pneumatic (Nosten©) devices (continuous monitoring of tracheal cuff pressure), in critically intubated children. This study aims to determine the effectiveness of the electronic device in the continuous monitoring of tracheal cuff pressure.

ELIGIBILITY:
Inclusion Criteria:

* Infants and children more than 2 days after birth at term and less than 5 years of age
* Patient intubated in the PICU with a cuffed endotracheal tube
* Predicted duration of mechanical ventilation > or = 24-hours
* Signed informed consent

Exclusion Criteria:

* Intubated with an uncuffed endotracheal tube
* Children admitted to the PICU with a previous tracheostomy
* Preterm children or infants less than 2 days post-term
* Patient under block neuromuscular treatment
* Patient enrolled in another trial that might influence this study results

Ages: 2 Days to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2021-04-16 (Actual); Study Completion 2021-04-16 (Actual)

PRIMARY OUTCOMES:
Percentage of time spend with over or under-inflation of the tracheal cuff | 12 hours
  Continuous recording of cuff pressure will be performed during the two 12-hours periods (electronic and pneumatic devices). The period was speared by a time of wash-out of 30 minutes

SECONDARY OUTCOMES:
The response time to a significant variation in cuff pressure | 12 hours
  Continuous recording of cuff pressure will be performed during the two 12-hours periods (electronic and pneumatic devices). Automated analysis of the response time in milliseconds to a change in cuff pressure of at least 15% above or below the target value

CONTACTS AND LOCATIONS:
Overall Officials: Boris LACARRA, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Stephane DAUGER, MD PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Robert Debré hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No